## Effects of Connectivity-based rTMS and State-Dependency on Amygdala Activation

NCT03746405

Statistical Plan

Date of Approval: February 14th, 2019

To examine whether active rTMS is more effective than sham rTMS to modulate amygdala activation, a repeated measure analysis of variance (ANOVA) will be performed on group data.

Prior to hypothesis testing, functional data will be preprocessed using FSL to remove noise and artifacts. Images will be normalized to a template, motion-corrected, high-pass filtered, and spatially smoothed (8 mm FWHM). Functional activations while subjects will be viewing fearful and neutral faces will be analyzed using standard procedures in FSL. The effects of stimulation (active vs. sham) and time (pre vs. post) will be compared on task-related functional activations. Activations will be considered significant at p < 0.05 with a minimum cluster extent threshold of 5 contiguous voxels. The same ANOVA will be performed on resting state and diffusion tensor imaging acquisitions. Participants with > 3 mm of movement during the acquisitions, will be excluded from the analyses